CLINICAL TRIAL: NCT02790411
Title: Adjustment Exploratory Protocols (MagnetoEncephaloGraphy Study : MEG, ElectroEncephaloGram : EEG, Magnetic Resonance Imaging : MRI, Functional MRI : MRIf, Motor Platform) and Functional Evaluation of New Non Invasive Devices (REX BIONICS Exoskeleton) in Healthy Volunteers
Brief Title: Adjustment Exploratory Protocols and Functional Evaluation of New Non Invasive Devices in Healthy Volunteers
Acronym: MAP-EFNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MAP-EFNI
Record Dates: First submitted 2016-05-12; First posted 2016-06-03 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Experimental): Imaging devices New Non Invasive Devices
  Interventions: Device: Imaging devices; Device: New Non Invasive Devices

INTERVENTIONS:
Device: Imaging devices — technological adjustment tests
Device: New Non Invasive Devices — Tests with REX BIONICS Exoskeleton

SUMMARY:
Parameters, sequences or paradigms optimisation in view of data quality and relevancy improvement.

DETAILED DESCRIPTION:
Various tests are needed for methodological optimization of the several devices (per-operative MRI, MEG, EEG, SPECT-CT, motor platform) of the technological platform.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Male or female aged over 18 years
* Registered in the French social security scheme
* Signed informed consent

Exclusion Criteria:

* Contraindication to Magnetoencephalography (MEG) and/or Electroencephalography (EEG)
* Contraindication to Magnetic resonance imaging (MRI)
* All categories of protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Magnetic brain activity | 2 hours
  MEG records
Brain imaging | 2 hours
  MRI and SPECT-CT records
Electrical brain activity | 2 hours
  EEG records
Motor activity parameters | 2 hours
  Motor platform records

CONTACTS AND LOCATIONS:
Locations (1):
- CLINATEC, Grenoble, France

IPD SHARING:
Plan to Share IPD: No